CLINICAL TRIAL: NCT01568697
Title: Oral Microbial and Immunological Characterization of Patients With Immune Dysfunction
Brief Title: Oral Bacteria and Immune System Problems Involved in Gum Disease (Periodontitis)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120100; 12-D-0100
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-21

CONDITIONS: Immunosuppression; Periodontal Disease; Healthy Subjects; Healthy Volunteer
Keywords: Microbiome; Periodontitis; Oral Mucosal Immunity; Oral Infection; Natural History; Immune Disorder; Periodontal Disease; Gum Disease; Healthy Volunteer; HV
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Immune System Diseases; Gingival Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy volunteers (with/without periodontal disease)
- Immune deficient patients: Subjects with known genetic immune deficiency
- Subjects with severe periodontitis of suspected genetic etiology and their family: Subjects with severe periodontitis of suspected genetic etiology and their family members

SUMMARY:
Background:

- Gum disease is a condition in which the tissue around the tooth root becomes swollen and infected. This condition can cause tooth loss if it is not treated. Who gets gum disease and how bad it will be depends on (1) the different bacteria in the mouth and (2) how the immune system of an individual handles these bacteria. Researchers want to look at the oral bacteria and genetic immune problems of different people to learn how these affect gum disease and other conditions of the mouth.

Objectives:

- To study how immune system problems may lead to problems in the mouth, including gum disease.

Eligibility:

* Children and adults at least 7 years of age who have genetic problems with their immune system.
* Healthy adults that have periodontal disease
* Health adults that do not have periodontal disease

Design:

* This study will involve a screening visit and a study visit.
* Participants will be screened with a medical history, blood work and a full oral and dental exam, including dental x-rays and photos.
* The study visit will involve collection of blood, urine, and other samples, including saliva, plaque, and gum swabs. Any abnormal tissue will sampled for a biopsy. Additional oral and dental exams will be performed. Participants will also answer questions about any current medical or dental problems.

DETAILED DESCRIPTION:
This is a cross sectional/natural history protocol designed to investigate the clinical,

microbiologic, and immunologic consequences of genetic immune defects in the oral cavity. The hypothesis is that genetic immune defects will lead to alterations in the local immune response and microbial colonization and ultimately predispose to susceptibility to oral infections and inflammatory conditions.

In the cross-sectional phase the following individuals will be enrolled, evaluated and screened for presence and severity of periodontitis, presence of a genetic defects and sampled for studies in oral immunity and microbiome: 1) individuals diagnosed with genetic immune defects 2) individuals with severe periodontitis of suspected genetic etiology and their family members 3) healthy volunteers. Subjects identified with a genetic immune defect and with presence of oral disease (primarily periodontitis) may enter the natural history phase of the study to be clinically followed at the National Institutes of Health (NIH) over time. This protocol aims to determine whether specific genetic immune defects will predispose to oral disease (primarily periodontitis) and to better understand consequences of immune deficiency on the oral immune response and microbiome.

Primary Objectives

1. Investigate the degree, scope, etiology and natural history of oral manifestations in patients with genetic immune defects.
2. Characterize the immune response in the oral cavity of patients with genetic immune defects.
3. Characterize the microbiome in the oral cavity of patients with genetic immune defects.

Secondary Objectives

1. Assay development/validation for the study of tissue immunity and microbiome characterization
2. Establishment of normative values for immune mediators and microbial elements at the oral cavity

Study Population (s)

The study population will include:

1. Subjects with genetic immune defects
2. Subjects with severe periodontitis of suspected genetic etiology and their family members
3. Healthy volunteers (with/without periodontal disease)

Design

This is a cross-sectional/natural history study for the evaluation of clinical, immunologic, and microbiologic oral manifestations (primarily periodontitis) in patients diagnosed with genetic immune defects or those with severe periodontitis of suspected genetic etiology and healthy volunteer subjects.

Cross Sectional Phase: Three groups of subjects will be enrolled in the cross-sectional phase of the study 1) individuals diagnosed with genetic immune defects 2) individuals with severe periodontitis of suspected genetic etiology and their family members that include parents or siblings 3) healthy volunteers (with/without periodontal disease). All groups will be evaluated for oral disease (periodontitis) may be and sampled for oral immunity, systemic immunity and microbiome characterization. Individuals with severe periodontitis in the presence/absence of a genetic defect may be offered the option of receiving standard of care inflammatory control periodontal treatment at NIH without travel compensation, following the cross-sectional portion of the study. Family members (parents or siblings) of individuals with periodontal disease of suspected genetic may be asked to participate in this study. During the course of genetic testing, family members may be enrolled in the cross sectional phase of the study for phenotyping and genetic testing.

Natural History Phase: Subjects identified with a genetic defect with the presence of oral disease may enroll in the natural history phase of the study to be followed clinically over time.

Primary Outcome Measures

1. Clinical intraoral characterization (i.e., presence and severity of periodontitis).
2. Characterize the immune response in the oral cavity of patients with genetic immune defects
3. Characterize the microbiome in the oral cavity of patients with genetic immune defects

Secondary Outcome Measures

1. Assay development/validation for the study of tissue immunity and microbiome characterization
2. Establishment of normative values for immune mediators and microbial elements at the oral cavity

Exploratory Outcome Measures

Initial data from this study may generate new hypotheses for investigation as part of this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with Genetic Immune Defects:

Patients with a known genetic immune defect will be eligible for screening inclusion under this protocol.

* Diagnosed with a genetic immune defect
* Willing to allow genetic testing

  * 7 years old

Subjects with Severe Periodontitis of Suspected Genetic Etiology:

* History of severe periodontitis prior to age <30
* Willing to allow genetic testing

  ->=7 years old
* In good general health

Family members of Subjects with Severe Periodontitis of Suspected Genetic Etiology:

-Willing to allow genetic testing

->=7 years old

Healthy Volunteer Subjects (with/without periodontitis):

* In good general health

  ->=18 years old
* Willing to allow genetic testing
* Have a minimum of 20 natural teeth

Inclusion Criteria for Natural History phase, all subjects:

* Diagnosis of genetic immune defect
* Presence of oral manifestation (primarily periodontitis)

Criteria for standard of care treatment:

* Active untreated disease (visible signs of tissue inflammation including erythema/edema, generalized bleeding upon probing)
* Periodontal disease defined as bone loss of >=5mm as measured on periodontal exam.

EXCLUSION CRITERIA:

All Subjects:

* History of Hepatitis B or C
* History of HIV
* Prior radiation therapy to the head or neck
* Have an active malignancy except localized basal or squamous cell carcinoma of the skin
* Have been treated with systemic chemotherapeutics or radiation therapy within 5 years of screening
* Pregnant or lactating
* If participation in the protocol would not be safe or in the subject s best interest in the opinion of either the PI or the primary medical team.

Additional Exclusions for Healthy Volunteers:

* Diagnosis of diabetes and/or HbA1C level >6%
* More than 3 hospitalizations in the last 3years
* Have an autoimmune disorder such as Lupus, Rheumatoid arthritis, etc.
* In the 3 months before study enrollment, have used any of the following:

  * Systemic (intravenous, intramuscular, or oral) antibiotics
  * Oral, intravenous, intramuscular, intranasal, or inhaled corticosteroids or other immunosuppressants (e.g., cyclosporine)
  * Cytokine therapy
  * Methotrexate or immunosuppressive chemotherapeutic agents
  * Large doses of commercial probiotics (>=10^8 colony-forming units or organisms per day); includes tablets, capsules, lozenges, chewing gum, or powders in which a probiotic is a primary component; ordinary dietary components such as fermented beverages/milks, yogurts, and foods do not apply
* Have used tobacco products (including e-cigarettes) within 1 year of screening
* Unwillingness to consent to oral biopsy
* NIH employees working in the Oral Immunity and Inflammation Unit and members of the Clinical Research Core Team will not be eligible for enrollment.

Additional Exclusions for Standard of Care Treatment at NIH:

* Mild/moderate non-active disease (absence of active inflammatory lesions)
* Subjects with urgent/complex restorative needs (ex. severe active carious lesions/fractured dentition)
* Subjects in need for advanced prosthetic needs (including implants and restorations)

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a cross sectional/natural history protocol designed to investigate the clinical, microbiologic, and immunologic consequences of genetic immune defects in the oral cavity. Three cohorts will be enrolled 1) subjects with genetic immune defects 2) subjects with severe periodontitis of suspected genetic etiology and their family members 3) healthy volunteers (with/without periodontal disease). The study involves detailed oral clinical and radiographic evaluations, standard laboratory testing and research sampling of blood and oral samples. All evaluations are performed at the NIH Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-10-05 (Actual)

PRIMARY OUTCOMES:
3. Characterize the microbiome in the oral cavity of patients with genetic immune defects | 25 years
  The primary clinical endpoints of the study are severity and types of oral disease: specifically for periodontal disease, mean PD, mean CAL, proportion of sites with PD >5 mm, and proportion of subjects with BOP, proportion of patient with other inflammatory conditions or infections of the oral cavity by immune disorder.Characterization of the oral microbiome in patients with monogenic immune defects. Immunologic endpoints: types and levels of immune mediators in the saliva, GCF, oral tissues, and/or blood.
2. Characterize the immune response in the oral cavity of patients with genetic immune defects | 25 years
  The primary clinical endpoints of the study are severity and types of oral disease: specifically for periodontal disease, mean PD, mean CAL, proportion of sites with PD >5 mm, and proportion of subjects with BOP, proportion of patient with other inflammatory conditions or infections of the oral cavity by immune disorder.Characterization of the oral microbiome in patients with monogenic immune defects. Immunologic endpoints: types and levels of immune mediators in the saliva, GCF, oral tissues, and/or blood.
1. Clinical intraoral characterization (i.e., presence and severity of periodontitis). | 25 years
  The primary clinical endpoints of the study are severity and types of oral disease: specifically for periodontal disease, mean PD, mean CAL, proportion of sites with PD >5 mm, and proportion of subjects with BOP, proportion of patient with other inflammatory conditions or infections of the oral cavity by immune disorder.Characterization of the oral microbiome in patients with monogenic immune defects. Immunologic endpoints: types and levels of immune mediators in the saliva, GCF, oral tissues, and/or blood.

SECONDARY OUTCOMES:
2. Establishment of normative values for immune mediators and microbial elements at the oral cavity | 25 years
  Validate methodologies for measuring levels of immune mediators in oral fluids - Establish normative values of immune mediators in oral fluids and tissues - Assay development; Develop new methodologies to study pathways of the immune response in the oral cavity - Assay development: Develop new methodologies to study the microbiome in the oral cavity
1. Assay development/validation for the study of tissue immunity and microbiome characterization | 25 years
  Validate methodologies for measuring levels of immune mediators in oral fluids - Establish normative values of immune mediators in oral fluids and tissues - Assay development; Develop new methodologies to study pathways of the immune response in the oral cavity - Assay development: Develop new methodologies to study the microbiome in the oral cavity

CONTACTS AND LOCATIONS:
Overall Officials: Niki M Moutsopoulos, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rescigno M. The intestinal epithelial barrier in the control of homeostasis and immunity. Trends Immunol. 2011 Jun;32(6):256-64. doi: 10.1016/j.it.2011.04.003. Epub 2011 May 11. PMID 21565554
- [Background] Novak N, Haberstok J, Bieber T, Allam JP. The immune privilege of the oral mucosa. Trends Mol Med. 2008 May;14(5):191-8. doi: 10.1016/j.molmed.2008.03.001. Epub 2008 Apr 7. PMID 18396104
- [Background] Maslowski KM, Mackay CR. Diet, gut microbiota and immune responses. Nat Immunol. 2011 Jan;12(1):5-9. doi: 10.1038/ni0111-5. PMID 21169997
- [Derived] Williams DW, Greenwell-Wild T, Brenchley L, Dutzan N, Overmiller A, Sawaya AP, Webb S, Martin D; NIDCD/NIDCR Genomics and Computational Biology Core; Hajishengallis G, Divaris K, Morasso M, Haniffa M, Moutsopoulos NM. Human oral mucosa cell atlas reveals a stromal-neutrophil axis regulating tissue immunity. Cell. 2021 Jul 22;184(15):4090-4104.e15. doi: 10.1016/j.cell.2021.05.013. Epub 2021 Jun 14. PMID 34129837
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-D-0100.html